CLINICAL TRIAL: NCT05699369
Title: A Cluster Randomised Controlled Trial to Evaluate the Effectiveness of Digital Health Interventions in Improving Non-communicable Disease Management During the Pandemic in Rural Pakistan
Brief Title: Interventions to Improve Non-communicable Disease Management During the Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Association for Social Development, Pakistan (Unknown); Canadian Institutes of Health Reesearch (Unknown)
Responsible Party: Principal Investigator, Xiaolin Wei, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRCT202112
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Noncommunicable Diseases; COVID-19
Keywords: digital health interventions; non-communicable diseases; cluster randomised trial; implementation science; resilience; Pakistan
MeSH Terms: conditions — Noncommunicable Diseases; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research team will mask the statisticians when data is presented and analyzed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): A comprehensive package of digital health interventions to connect patients, patient champions and public health providers to improve the management of non-communicable diseases (NCDs) during the pandemic will be implemented, including 1) providing training to health providers regarding an integrated NCD-COVID guideline; 2) using a smartphone app to improve NCD case management and linking with patient champions; and 3) employing telementoring platform to improve quality of care. Patient champions are experienced patients who can provide peer support.
  Interventions: Other: Digital health interventions
- Control arm (No Intervention): Usual care, which is routine hypertension and diabetes diagnosis and treatment under the World Diabetes Foundation (WDF) project will be implemented. The WDF project provides initial Zoom-based training of NCD care to rural health center (RHC) staff, but no tele-mentorship is offered. Under the usual care, patients with hypertension or diabetes are required to visit RHCs every month to renew their medications and measure their blood pressure. No other interventional components will be implemented in the control arm.

INTERVENTIONS:
Other: Digital health interventions — Described in arm descriptions.
  Arms: Intervention arm

SUMMARY:
This randomized controlled trial aims to implement and evaluate a comprehensive package of digital health interventions for integrated COVID-non-communicable diseases (NCDs) care to manage NCDs in primary care facilities in rural Pakistan. The main questions it aims to answer are 1) whether such interventions are effective; 2) how they were implemented; and 3) whether such interventions are cost-effective.

30 rural health centers in Punjab Province, Pakistan will be randomized into two groups. The intervention group will provide a comprehensive package of digital health interventions to connect patients, patient champions, and public health providers to improve the management of NCDs during the pandemic, including 1) providing training to health providers regarding an integrated NCD-COVID guideline; 2) using a smartphone app to improve NCD case management and linking with patient champions; and 3) employing telementoring platform to improve quality of care. Usual care will be provided in the control group. Researchers will compare the two groups to see if the systolic blood pressure can be controlled better in the intervention group at 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the catchment of selected rural health centers;
* Provide informed consent;
* Newly diagnosed of hypertension, i.e., having a baseline blood pressure reading (recorded from the second blood pressure reading using a validated electronic blood pressure machine) of more than 140/90 mmHg; or who is an existing hypertensive patient but with uncontrolled blood pressure with a baseline blood pressure over 140/90 mmHg;
* Have a smartphone or can access a smartphone from a relative.

Exclusion Criteria:

* Patients having an acute cardiovascular event in the last three months, terminal disease, or other conditions that the rural health center staff determine that will make participation impossible.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (mmHg) measured in the rural health center | At 10 months

SECONDARY OUTCOMES:
Diastolic blood pressure (mmHg) measured in the rural health center | At 10 months
Percentage of patients with controlled blood pressure measured below 140/90 mmHg for patients with hypertension but without diabetes, and below 130/80 mmHg for patients with diabetes | At 10 months
Random blood glucose (mmol/L) | At 10 months
Body mass index (BMI) | At 10 months
Number of consultations with RHC doctors, including both in-person and virtual consultations | During the 10-month intervention period
Systolic and diastolic blood pressure | At 6 months
Proportion of patients who have had at least three doses of COVID vaccinations | At 10 months
Proportion of participants been admitted to district hospitals for any reasons | During the 10-month intervention period
All-cause mortality rate | During the 10-month intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Wei, PhD, Principal Investigator — University of Toronto
Locations (1):
- Primary care facilities, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
According to the ethical agreements, the data is only available for research purpose of the study team. Individual patient data cannot be posted and downloaded in a public data depository. Anonymous data can be shared upon request to the study contacts with joint ethics application to the University of Toronto.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication in peer-reviewed journals.
Access Criteria: The research team will aim to publish them in open access journals as priority so that all other researchers will freely access to them.

REFERENCES:
- [Derived] Wei X, Khan N, Durrani H, Muzaffar N, Haldane V, Walley JD, Thorpe K, Ge E, Ge S, Dodd W, Wallace J, Aslanyan G, Laporte A, Khan MA. Protocol for a pragmatic cluster randomised controlled trial to evaluate the effectiveness of digital health interventions in improving non-communicable disease management during the pandemic in rural Pakistan. PLoS One. 2023 Oct 10;18(10):e0282543. doi: 10.1371/journal.pone.0282543. eCollection 2023. PMID 37816010